CLINICAL TRIAL: NCT00950807
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Way Cross-Over Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of GSK573719 Administered Once- and Twice-Daily in Subjects With COPD
Brief Title: GSK573719 Dose Ranging Study in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113073
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Dose ranging; Chronic Bronchitis; Long-acting muscarinic antagonist; cross-over; COPD; Emphysema; Chronic Obstructive Pulmonary Disease (COPD); anticholinergic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Tiotropium (Active Comparator): Tiotropium
  Interventions: Drug: Tiotropium
- Arm 1 (Experimental): GSK573719 1000mcg once daily
  Interventions: Drug: GSK573179
- Arm 2 (Experimental): GSK573719 500mcg once daily
  Interventions: Drug: GSK573179
- Arm 3 (Experimental): GSK573719 250mcg once daily
  Interventions: Drug: GSK573179
- Arm 4 (Experimental): GSK573719 125mcg once daily
  Interventions: Drug: GSK573179
- Arm 5 (Experimental): GSK573719 62.5 mcg once daily
  Interventions: Drug: GSK573179
- Arm 6 (Experimental): GSK573719 250mcg twice daily
  Interventions: Drug: GSK573179
- Arm 7 (Experimental): GSK573719 125mcg twice daily
  Interventions: Drug: GSK573179
- Arm 8 (Experimental): GSK573719 62.5mcg twice daily
  Interventions: Drug: GSK573179

INTERVENTIONS:
Drug: Tiotropium — long-acting muscarinic receptor antagonist; 18mcg once-daily
  Arms: Tiotropium
Drug: Placebo — Inactive/ excipients only
  Arms: Placebo
Drug: GSK573179 — GSK573179 investigational drug
  Arms: Arm 1; Arm 2; Arm 3; Arm 4; Arm 5; Arm 6; Arm 7; Arm 8

SUMMARY:
The study will evaluate the dose response, safety, and pharmacokinetics of GSK573719 compared with placebo in subjects with COPD.

DETAILED DESCRIPTION:
This is multicenter, randomized, double-blind, double-dummy, placebo-controlled, three-way cross-over, incomplete block design study to evaluation of 5 doses of GSK573719 administered once-daily and 3 doses of GSK573719 administered twice-daily over 14 days in subjects with COPD and will include tiotropium as an open-label active control. The pharmacokinetic profile of GSK573719 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated written informed consent prior to study participation
* Males or females of non-childbearing potential
* 40 to 80 years of age
* COPD diagnosis
* 10 pack-years history or greater of cigarette smoking
* Post-bronchodilator FEV1/FVC ratio of 0.70 or less
* Post-bronchodilator FEV1 of 35 to 70% of predicted normal

Exclusion Criteria:

* Asthma
* Other significant respiratory disorders besides COPD, including alpha-1 deficiency
* Previous lung resection surgery
* Use of oral steroids or antibiotics for a COPD exacerbation within 6 weeks of screening
* Hospitalization for COPD or pneumonia within 3 months of screening
* Any significant disease that would put subject at risk through study participation
* BMI greater than 35
* Pacemaker
* Significantly abnormal ECG, Holter, or clinical lab finding (including Hepatitis B or C)
* Cancer
* Allergy or hypersensitivity to anticholinergics or inhaler excipients
* Diseases that would contra-indicate the use of anticholinergics
* Use of oral corticosteroids within 6 weeks of screening
* Use of long-acting beta-agonists within 48 hours of screening
* Use of tiotropium within 14 days of screening
* Use of theophyllines or anti-leukotrienes within 48 hours of screening
* Use of short-acting bronchodilators within 4 to 6 hours of screening
* Use of investigational medicines within 30 days of screening
* Use of high dose inhaled corticosteroids
* Use of long-term oxygen therapy, CPAP or NIPPV
* Previous use of GSK573719

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2009-09-01; Primary Completion 2010-03-01 (Actual); Study Completion 2010-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- United States (10):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
- Germany (8):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Donohue JF, Anzueto A, Brooks J, Mehta R, Kalberg C, Crater G. A randomized, double-blind dose-ranging study of the novel LAMA GSK573719 in patients with COPD. Respir Med. 2012 Jul;106(7):970-9. doi: 10.1016/j.rmed.2012.03.012. Epub 2012 Apr 10. PMID 22498110
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113073 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who were eligible completed a 4- to 7-day Run-in period prior to randomization. The treatment (trt) phase was comprised of three 14-day trt periods. Par. were randomly assigned to receive a sequence of placebo and 2 of the 9 active trts over the trt phase. Participant Flow data are presented by treatment rather than sequence.
Groups:
- Placebo: Participants received matching placebo in the morning via dry powder inhaler (DPI) A and in the evening via DPI B for 14 days.
- UMEC 62.5 µg QD: Participants received umeclidinium bromide (UMEC) 62.5 micrograms (µg) in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 125 µg QD: Participants received UMEC 125 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 250 µg QD: Participants received UMEC 250 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 500 µg QD: Participants received UMEC 500 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 1000 µg QD: Participants received UMEC 1000 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- UMEC 62.5 µg BID: Participants received UMEC 62.5 µg in the morning via DPI A and in the evening via DPI B for 14 days.
- UMEC 125 µg BID: Participants received UMEC 125 µg in the morning via DPI A and in the evening via DPI B for 14 days.
- UMEC 250 µg BID: Participants received UMEC 250 µg in the morning via DPI A and in the evening via DPI B for 14 days.
- Tiotropium 18 µg QD: Participants received tiotropium bromide 18 µg in the morning via the HandiHaler and placebo in the evening via DPI B for 14 days.
Period: Treatment Period 1
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 500 µg QD | UMEC 1000 µg QD | UMEC 62.5 µg BID | UMEC 125 µg BID | UMEC 250 µg BID | Tiotropium 18 µg QD
Started | 59 | 13 | 14 | 12 | 13 | 13 | 12 | 14 | 13 | 13
Completed | 56 | 13 | 13 | 12 | 12 | 11 | 12 | 14 | 12 | 13
Not Completed | 3 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 500 µg QD | UMEC 1000 µg QD | UMEC 62.5 µg BID | UMEC 125 µg BID | UMEC 250 µg BID | Tiotropium 18 µg QD
Started | 56 | 13 | 13 | 12 | 12 | 11 | 12 | 14 | 12 | 13
Completed | 51 (Participants withdrawing during washout are counted under the last treatment taken.) | 13 (Participants withdrawing during washout are counted under the last treatment taken.) | 13 (Participants withdrawing during washout are counted under the last treatment taken.) | 11 (Participants withdrawing during washout are counted under the last treatment taken.) | 11 (Participants withdrawing during washout are counted under the last treatment taken.) | 11 (Participants withdrawing during washout are counted under the last treatment taken.) | 10 (Participants withdrawing during washout are counted under the last treatment taken.) | 13 (Participants withdrawing during washout are counted under the last treatment taken.) | 11 (Participants withdrawing during washout are counted under the last treatment taken.) | 13 (Participants withdrawing during washout are counted under the last treatment taken.)
Not Completed | 5 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol-defined Stopping Criteria | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 500 µg QD | UMEC 1000 µg QD | UMEC 62.5 µg BID | UMEC 125 µg BID | UMEC 250 µg BID | Tiotropium 18 µg QD
Started | 53 (By crossover design, participants were assigned to a different treatment arm in each period.) | 13 (By crossover design, participants were assigned to a different treatment arm in each period.) | 10 (By crossover design, participants were assigned to a different treatment arm in each period.) | 13 (By crossover design, participants were assigned to a different treatment arm in each period.) | 13 (By crossover design, participants were assigned to a different treatment arm in each period.) | 10 (By crossover design, participants were assigned to a different treatment arm in each period.) | 10 (By crossover design, participants were assigned to a different treatment arm in each period.) | 13 (By crossover design, participants were assigned to a different treatment arm in each period.) | 11 (By crossover design, participants were assigned to a different treatment arm in each period.) | 11 (By crossover design, participants were assigned to a different treatment arm in each period.)
Completed | 51 | 12 | 10 | 12 | 13 | 9 | 9 | 10 | 11 | 11
Not Completed | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Protocol-defined Stopping Criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Period: Washout Period 2
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 500 µg QD | UMEC 1000 µg QD | UMEC 62.5 µg BID | UMEC 125 µg BID | UMEC 250 µg BID | Tiotropium 18 µg QD
Started | 51 | 12 | 10 | 12 | 13 | 9 | 9 | 10 | 11 | 11
Completed | 47 (Participants withdrawing during washout are counted under the last treatment taken.) | 11 (Participants withdrawing during washout are counted under the last treatment taken.) | 10 (Participants withdrawing during washout are counted under the last treatment taken.) | 11 (Participants withdrawing during washout are counted under the last treatment taken.) | 12 (Participants withdrawing during washout are counted under the last treatment taken.) | 9 (Participants withdrawing during washout are counted under the last treatment taken.) | 8 (Participants withdrawing during washout are counted under the last treatment taken.) | 9 (Participants withdrawing during washout are counted under the last treatment taken.) | 11 (Participants withdrawing during washout are counted under the last treatment taken.) | 11 (Participants withdrawing during washout are counted under the last treatment taken.)
Not Completed | 4 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol-defined Stopping Criteria | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 500 µg QD | UMEC 1000 µg QD | UMEC 62.5 µg BID | UMEC 125 µg BID | UMEC 250 µg BID | Tiotropium 18 µg QD
Started | 46 (By crossover design, participants were assigned to a different treatment arm in each period.) | 9 (By crossover design, participants were assigned to a different treatment arm in each period.) | 10 (By crossover design, participants were assigned to a different treatment arm in each period.) | 11 (By crossover design, participants were assigned to a different treatment arm in each period.) | 12 (By crossover design, participants were assigned to a different treatment arm in each period.) | 9 (By crossover design, participants were assigned to a different treatment arm in each period.) | 12 (By crossover design, participants were assigned to a different treatment arm in each period.) | 10 (By crossover design, participants were assigned to a different treatment arm in each period.) | 9 (By crossover design, participants were assigned to a different treatment arm in each period.) | 11 (By crossover design, participants were assigned to a different treatment arm in each period.)
Completed | 45 | 9 | 10 | 11 | 12 | 9 | 11 | 9 | 9 | 10
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol-defined Stopping Criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Treatments: The treatment phase was comprised of three 14-day treatment periods, each separated by a 10-14 day washout period. Participants were randomly assigned to receive a sequence of placebo and 2 of the 9 active treatments :
  UMEC 62.5, 125, 250, 500, and 1000 µg QD, UMEC 62.5, 125, and 250 µg BID, tiotropium 18 µg QD.
Arm/Group | All Study Treatments
Number analyzed (Participants) | 176
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 101
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 4
  White | 172

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Day 15 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Treatment Day 15 is defined as the value obtained 24 hours after the morning dose administered on Day 14. Analysis were performed using a mixed model with covariates of mean Baseline, period Baseline, treatment and period as fixed effects and participant as a random effect. Baseline is the FEV1 value recorded pre-dose on Day 1 of each treatment period; mean Baseline is the mean of the Baselines for each participant and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Change from Baseline for each treatment period is the trough FEV1 at Day 15 minus the Baseline value for that treatment period.
Time Frame: Baseline and Day 15 of each treatment period (up to Study Day 71)
Population: Modified Intent-To-Treat (mITT) Population: all participants randomized to treatment who received at least one dose of study medication. All participants with >=1 post-baseline assessment and non-missing covariate data are included in the analysis. The number of participants represents participants who provided data at Day 15.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- UMEC 62.5 µg QD: Participants received UMEC 62.5 µg in the morning via DPI A and placebo in the evening via DPI B for 14 days.
- Tio 18 µg QD: Participants received tiotropium bromide 18 µg in the morning via the HandiHaler and placebo in the evening via DPI B for 14 days.
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 500 µg QD | UMEC 1000 µg QD | UMEC 62.5 µg BID | UMEC 125 µg BID | UMEC 250 µg BID | Tio 18 µg QD
Number analyzed (Participants) | 150 | 34 | 33 | 35 | 37 | 29 | 31 | 33 | 32 | 34
Liters | -0.047 (0.017) | 0.081 (0.033) | 0.099 (0.034) | 0.048 (0.033) | 0.092 (0.032) | 0.138 (0.036) | 0.032 (0.035) | 0.087 (0.034) | 0.124 (0.034) | 0.058 (0.033)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.128, 95% CI 2-sided [0.060 to 0.196]
Statistical Analysis 2: Comparison: Placebo vs UMEC 125 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.147, 95% CI 2-sided [0.077 to 0.216]
Statistical Analysis 3: Comparison: Placebo vs UMEC 250 µg QD; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = 0.095, 95% CI 2-sided [0.027 to 0.162]
Statistical Analysis 4: Comparison: Placebo vs UMEC 500 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.140, 95% CI 2-sided [0.074 to 0.205]
Statistical Analysis 5: Comparison: Placebo vs UMEC 1000 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.186, 95% CI 2-sided [0.113 to 0.259]
Statistical Analysis 6: Comparison: Placebo vs UMEC 62.5 µg BID; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [0.008 to 0.151]
Statistical Analysis 7: Comparison: Placebo vs UMEC 125 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.134, 95% CI 2-sided [0.064 to 0.204]
Statistical Analysis 8: Comparison: Placebo vs UMEC 250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.172, 95% CI 2-sided [0.101 to 0.242]
Statistical Analysis 9: Comparison: Placebo vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = 0.105, 95% CI 2-sided [0.037 to 0.173]

2. Secondary Outcome: Change From Baseline (BL) in Weighted Mean FEV1 Over 0 to 24 Hours Obtained Post-dose on Day 14 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The weighted mean FEV1 was calculated using 0-24 hour (h) post-dose measurements at Day 14 of each treatment period, which included pre-dose and post-dose 1, 3, 6, 9, 12, 13, 15, 18, 21 and 24 hours. Analysis performed using a mixed model with covariates mean BL, period BL, treatment and period as fixed effects and participant as a random effect. BL is the FEV1 value recorded pre-dose on Day 1 of each TP; mean BL is the mean of the BLs for each participant and period BL is the difference between the BL and the mean BL in each TP for each participant. Change from BL for each TP is the trough FEV1 at Day 15 minus the BL value for that TP.
Time Frame: Baseline and Day 14 of each treatment period (TP; up to Study Day 70)
Population: mITT Population. All participants with >=1 post-Baseline assessment and non-missing covariate data are included in the analysis. The number of participants represents participants who provided data at Day 14.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 500 µg QD | UMEC 1000 µg QD | UMEC 62.5 µg BID | UMEC 125 µg BID | UMEC 250 µg BID | Tio 18 µg QD
Number analyzed (Participants) | 143 | 33 | 33 | 34 | 36 | 29 | 30 | 32 | 31 | 33
Liters | -0.059 (0.014) | 0.085 (0.025) | 0.077 (0.025) | 0.077 (0.025) | 0.072 (0.024) | 0.080 (0.027) | 0.062 (0.026) | 0.083 (0.025) | 0.075 (0.026) | 0.069 (0.025)

3. Secondary Outcome: Change From Baseline (BL) in Serial FEV1 Over 0-28 Hours After the Morning Dose at Day 14 of Each Treatment Period
Description: Serial FEV1 for OQ dosing is recorded at the pre-AM dose (time 0 h) and at 1, 3, 6, 9, 12,13, 15, 18, 21, 24 and 28 hs after the AM dose on D 14. For BID dosing, the 12 h AM dose corresponds to the pre-PM dose, 13 h AM dose corresponds to the 1 h PM dose, 15 h AM dose corresponds to the 3 h PM dose, 18 h AM corresponds to the 6 h PM dose, 21 h AM dose corresponds to 9 h PM dose, 24 h AM dose corresponds to the 12 h PM dose and 28 h AM dose corresponds to the 16 h PM dose in the table. Analysis performed using a mixed model with covariates of mean BL, period BL, trt, period, time, time by period BL interaction, time by mean BL interaction and time by trt interaction as fixed effects and par. as a random effect. BL is the FEV1 value recorded pre-dose on D 1 of each TP; mean BL is the mean of the BLs for each par. and period BL is the difference between the BL and the mean BL in each TP for each par. Change from BL for each TP is the trough FEV1 at Day 15 minus the BL value for that TP.
Time Frame: Baseline and Day (D) 14 of each treatment period (TP; up to Study Day 70)
Population: mITT Population. All par. with >=1 post-BL assessment and non-missing covariate data are included in the analysis. Different par. may have been analyzed at different time points (n=X, X, X, X in the category titles), so the overall number of par. analyzed reflects everyone in the mITT Population with data available at >=1 time point.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 500 µg QD | UMEC 1000 µg QD | UMEC 62.5 µg BID | UMEC 125 µg BID | UMEC 250 µg BID | Tio 18 µg QD
Number analyzed (Participants) | 152 | 34 | 33 | 35 | 37 | 30 | 32 | 33 | 32 | 34
Liters
  Pre-AM dose, n=152,34,33,35,37,30,32,33,32,34 | -0.002 (0.016) | 0.140 (0.031) | 0.101 (0.032) | 0.167 (0.031) | 0.095 (0.030) | 0.120 (0.033) | 0.096 (0.032) | 0.139 (0.032) | 0.152 (0.032) | 0.129 (0.031)
  1 hour AM, n=151,34,31,35,37,29,32,33,32,34 | 0.022 (0.018) | 0.246 (0.035) | 0.164 (0.037) | 0.140 (0.035) | 0.056 (0.034) | 0.072 (0.038) | 0.159 (0.037) | 0.132 (0.036) | 0.142 (0.037) | 0.229 (0.036)
  3 hour AM, n=150,34,32,35,37,29,31,33,32,34 | -0.003 (0.017) | 0.157 (0.034) | 0.158 (0.035) | 0.222 (0.034) | 0.142 (0.033) | 0.148 (0.037) | 0.153 (0.036) | 0.112 (0.035) | 0.153 (0.036) | 0.191 (0.035)
  6 hour AM, n=151,34,33,35,37,30,32,33,31,34 | -0.019 (0.016) | 0.137 (0.031) | 0.114 (0.032) | 0.149 (0.031) | 0.120 (0.030) | 0.105 (0.034) | 0.090 (0.033) | 0.100 (0.032) | 0.141 (0.033) | 0.152 (0.032)
  9 hour AM, n=149,33,33,34,37,30,31,32,32,33 | -0.033 (0.016) | 0.121 (0.033) | 0.077 (0.033) | 0.123 (0.032) | 0.118 (0.031) | 0.076 (0.035) | 0.105 (0.034) | 0.104 (0.033) | 0.099 (0.034) | 0.105 (0.033)
  12 hour AM, n=150,34,33,34,37,30,31,32,32,33 | -0.068 (0.018) | 0.087 (0.035) | 0.083 (0.036) | 0.084 (0.035) | 0.096 (0.034) | 0.074 (0.038) | 0.058 (0.037) | 0.099 (0.036) | 0.074 (0.036) | 0.153 (0.036)
  13 hour AM, n=147,33,33,35,37,29,31,33,32,33 | -0.082 (0.016) | 0.071 (0.031) | 0.077 (0.031) | 0.071 (0.031) | 0.103 (0.030) | 0.096 (0.033) | 0.066 (0.032) | 0.018 (0.032) | 0.048 (0.032) | 0.065 (0.031)
  15 hour AM, n=151,34,33,35,37,29,30,33,32,34 | -0.085 (0.016) | 0.074 (0.031) | 0.051 (0.032) | 0.069 (0.031) | 0.038 (0.030) | 0.050 (0.033) | 0.085 (0.033) | 0.054 (0.032) | 0.096 (0.032) | 0.036 (0.031)
  18 hour AM, n=148,33,33,35,36,29,31,33,32,34 | -0.145 (0.016) | -0.053 (0.033) | 0.002 (0.033) | -0.018 (0.032) | -0.007 (0.031) | 0.001 (0.035) | -0.020 (0.034) | 0.016 (0.033) | -0.048 (0.033) | -0.097 (0.032)
  21 hour AM, n=150,34,33,35,37,29,29,33,32,34 | -0.147 (0.017) | 0.009 (0.034) | 0.035 (0.034) | -0.036 (0.034) | 0.004 (0.033) | 0.006 (0.037) | -0.059 (0.036) | 0.029 (0.035) | -0.005 (0.035) | -0.060 (0.034)
  24 hour AM, n=150,34,33,35,37,29,31,33,32,34 | -0.051 (0.017) | 0.067 (0.033) | 0.093 (0.034) | 0.045 (0.033) | 0.088 (0.032) | 0.142 (0.036) | 0.021 (0.035) | 0.091 (0.034) | 0.139 (0.035) | 0.047 (0.033)
  28 hour AM, n=145,34,33,35,37,29,31,33,32,34 | 0.065 (0.018) | 0.179 (0.035) | 0.177 (0.036) | 0.212 (0.035) | 0.143 (0.034) | 0.191 (0.038) | 0.164 (0.037) | 0.219 (0.036) | 0.185 (0.037) | 0.108 (0.035)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication up to 10 weeks.
Description: On-treatment AEs and non-serious AEs are reported for members of the mITT Population, comprised of all participants who were randomized to treatment and who had received at least one dose of randomized study medication during treatment period.
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD | UMEC 250 µg QD | UMEC 500 µg QD | UMEC 1000 µg QD | UMEC 62.5 µg BID | UMEC 125 µg BID | UMEC 250 µg BID | Tio 18 µg QD
Serious Adverse Events (participants affected / at risk) | 0/158 | 0/35 | 0/34 | 2/36 | 0/38 | 0/32 | 0/34 | 1/37 | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 11/158 | 2/35 | 3/34 | 8/36 | 9/38 | 13/32 | 4/34 | 4/37 | 10/33 | 3/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | UMEC 62.5 µg QD (N=35) | UMEC 125 µg QD (N=34) | UMEC 250 µg QD (N=36) | UMEC 500 µg QD (N=38) | UMEC 1000 µg QD (N=32) | UMEC 62.5 µg BID (N=34) | UMEC 125 µg BID (N=37) | UMEC 250 µg BID (N=33) | Tio 18 µg QD (N=35)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | UMEC 62.5 µg QD (N=35) | UMEC 125 µg QD (N=34) | UMEC 250 µg QD (N=36) | UMEC 500 µg QD (N=38) | UMEC 1000 µg QD (N=32) | UMEC 62.5 µg BID (N=34) | UMEC 125 µg BID (N=37) | UMEC 250 µg BID (N=33) | Tio 18 µg QD (N=35)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 4 | 2 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 1 | 3 | 1 | 2 | 0 | 1 | 3 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 4 | 2 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.